CLINICAL TRIAL: NCT06058923
Title: Minimally Invasive Surgical Techniques of Single Versus Double-flap for the Treatment of Isolated Intrabony Defects: a Randomized Controlled Clinical Trial
Brief Title: MIST Versus M-MIST for the Treatment of Intrabony Defects
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Enilson Antonio Sallum, PhD, Chair of Periodontology Area, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69036023.5.0000.5418
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Periodontitis; Intrabony Periodontal Defect; Periodontitis, Chronic
MeSH Terms: conditions — Periodontitis; Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: Randomized controlled double-blind parallel-design clinical trial with a longitudinal duration of 12 months per participant, involving surgical therapeutic intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally Invasive Surgical Technique (MIST) (Active Comparator): Double flap minimally invasive surgery for the access of intrabony defects
  Interventions: Procedure: MIST
- Modified Minimally Invasive Surgical Technique (M-MIST) (Experimental): Single flap minimally invasive surgery for the access of intrabony defects
  Interventions: Procedure: M-MIST

INTERVENTIONS:
Procedure: M-MIST — This is characterized by a vestibular mucoperiosteal envelope flap without relaxing incisions. Sulcular incisions will be made on the vestibular surface of the teeth included in the surgical area, adjacent to the infraosseous defect. The mesiodistal extension of the flap will be kept to a minimum necessary to access the defect. In the papillary area over the infraosseous defect, an oblique or horizontal incision will be made at the level of the interdental papilla, following the contour of the bone crest. The vestibular flap will be elevated, leaving the lingual/palatal portion adhered, only to allow access to the bone defect. The defect will be instrumented with mini-curettes and specific ultrasonic tips, and the defect will be filled only with a blood clot after this procedure. Primary closure will be achieved with internal vertical and/or horizontal mattress sutures, which may be complemented with simple sutures, all using specific suture threads.
  Other Names: Minimally invasive single flap technique
  Arms: Modified Minimally Invasive Surgical Technique (M-MIST)
Procedure: MIST — A vestibular envelope flap, without vertical relaxing incisions, will be raised on the vestibular and lingual/palatal sides. Primary intrasulcular incisions will be made to the alveolar crest, encompassing the teeth included in the surgical area. In the interproximal area, incisions will follow the principle of preserving the papilla (Modified Papilla Preservation Technique = MPPT or Simplified Papilla Preservation Flap = SPPF), depending on the available interproximal space (Cortellini et al., 1995, 1999). The mesiodistal extension of the flap will be minimized to provide adequate access to the defect. The defect will be instrumented using mini-curettes and specific ultrasonic tips, and the defect will be filled only with a blood clot after these procedures. Flap closure will be achieved with internal horizontal and/or vertical mattress sutures, which may be modified or complemented with simple sutures, all using specific suture threads.
  Other Names: Minimally invasive double flap technique
  Arms: Minimally Invasive Surgical Technique (MIST)

SUMMARY:
This is a 12-month longitudinal, double-blind, parallel-design randomized controlled clinical trial involving surgical therapeutic intervention (Phase 4). It will include 50 participants aged 21 diagnosed with periodontitis (Stage III/IV, Grade A or B), divided into a Test Group (n=25, Minimally invasive single-flap surgery) and a Control Group (n=25, Minimally invasive double-flap surgery). The objective of this randomized, double-blind clinical study is to compare clinical, radiographic, and patient-centered outcomes between minimally invasive single-flap and double-flap techniques in treating isolated infra-bony defects. Twenty-five patients will be treated using the single-flap approach, and 25 patients will receive the double-flap elevation technique. Clinical parameters (plaque and bleeding scores, probing depth, gingival recession, clinical attachment level, and papillary dimensions), digital measurements (changes in gingival margin and papillary volume), radiographic assessments, and patient-centered outcomes (VAS scale) will be evaluated immediately before surgery, at 6 and 12 months post-procedure, while early healing will be assessed after 1 and 2 weeks following the procedures. Mean values and standard deviations will be calculated for each variable, normal distribution will be tested using the Shapiro-Wilk test, and comparisons will be conducted using Student's t-test and one-way ANOVA. A significance level of 5% will be used for all analyses.

DETAILED DESCRIPTION:
This is a clinical trial, a randomized controlled double-blind parallel-design study with a 12-month follow-up. Participants will be recruited from patients diagnosed with periodontitis (Stage III/IV, Grade A or B) based on inclusion and exclusion criteria at the Postgraduate Periodontics Clinic of the Dental College of Piracicaba in the State University of Campinas (FOP-UNICAMP). The sample size calculation was based on a previous study, resulting in 50 participants, with 25 in each group. Participants will be randomly assigned to two treatment groups: Control Group (double-flap minimally invasive surgery) and Test Group (single-flap minimally invasive surgery).

This study will include clinical, digital, radiographic and patient-related outcome measures parameters. Clinical parameters including plaque index, bleeding on probing, probing depth, gingival recession, clinical attachment level, and early healing index will be measured at baseline, 6 months, and 12 months. Digital parameters, including mean change in papillary volume (mmVP) and change in gingival margin (mGM), will be assessed through intraoral scanning at baseline and 12 months. Radiographic measurements (linear, angular, and subtraction) will be performed before surgery and 12 months after using specialized software. Patient perception of pain and analgesic consumption will be evaluated using the Visual Analogue Scale (VAS) at various time points post-surgery (1-14 days after surgical intervention).

The clinical protocol involves pre-surgical therapy, surgical therapy, and post-operative care. After recording all the parameters through periodontal evaluation, X-ray acquisition procedures and intraoral scanning, a full-mouth supra and subgingival scaling and root planing will be performed. Afterwards, the surgery will be performed, following the randomization. Patients will receive post-operative analgesics and instructions for oral hygiene modifications. Periodontal maintenance will occur at specific intervals after surgery (1 month after surgery, 2 months after surgery, 4 months after surgery, 7 months after surgery, 10 months after surgery and 12 months after surgery).

For the statistical analysis, descriptive statistics will be used, and normality will be tested. Comparisons will be made using Student's t-test, one-way ANOVA, or non-parametric tests if data do not follow a normal distribution. A significance level of 5% will be used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals
* Diagnosis of periodontitis (stage III/IV - grade A or B)
* Presence of 20 or more teeth in the oral cavity
* Presence of at least one isolated interproximal infra-bony defect (without extension of the defect to the lingual or palatal area - assessed with preoperative bone sounding), with a probing depth of 6 mm or more, and a radiographic infra-bony component ≥ 4 mm, not associated with bifurcation areas, in anterior or premolar teeth (Schincaglia et al., 2015)
* Plaque index and bleeding on probing index ≤ 20% (baseline)
* Individuals providing informed and voluntary consent

Exclusion Criteria:

* Individuals who are not available for study evaluation appointments
* Systemic conditions that contraindicate periodontal surgery
* Patients requiring prophylactic antibiotics
* Compromised systemic condition (leukocyte dysfunction, bleeding disorders, neoplasms, uncontrolled metabolic or endocrine disorders, HIV infection)
* Individuals using bisphosphonates (oral or injectable use)
* Individuals using antibiotics and steroids (within 6 months prior to the study start)
* Illicit drug users
* Smokers
* Individuals with the tooth associated with the infra-bony defect having inadequate restoration, endodontic lesion, inadequate endodontic treatment, untreated carious lesions, and Grade III mobility
* Pregnant and lactating Women

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Probing Depth | 6 months and 1 year
  Reduction of Probing Depth

SECONDARY OUTCOMES:
Clinical Attachment Level | 6 months and 1 year
  Gain of the Clinical Attachment Level
Subtraction Radiography | 1 year
  Gain of bone level

CONTACTS AND LOCATIONS:
Overall Officials: Thais FM Paschoal, MsC, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Piracicaba Dental School, State University of Campinas, Piracicaba, São Paulo, Brazil